CLINICAL TRIAL: NCT00880087
Title: Therapeutic Hypothermia After Pediatric Cardiac Arrest (In Hospital)
Brief Title: Therapeutic Hypothermia to Improve Survival After Cardiac Arrest in Pediatric Patients-THAPCA-IH [In Hospital] Trial
Acronym: THAPCA-IH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Frank W. Moler, M.D, M.S, Professor of Pediatrics, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 620; U01HL094345 (NIH)
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Results first posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-05

CONDITIONS: Cardiac Arrest
Keywords: Cardiac Arrest; Cardiopulmonary Arrest; Pediatric Cardiac Arrest; VABS; Vineland Adaptive Behavior Scale; POPC/PCPC; hypoxic-ischemic encephalopathy
MeSH Terms: conditions — Heart Arrest; Hypoxia-Ischemia, Brain | interventions — Hypothermia, Induced

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Therapeutic Hypothermia (Experimental): Participants will receive therapeutic hypothermia after experiencing cardiac arrest.
  Interventions: Procedure: Therapeutic Hypothermia
- Therapeutic Normothermia (Active Comparator): Participants will receive therapeutic normothermia after experiencing cardiac arrest.
  Interventions: Procedure: Therapeutic Normothermia

INTERVENTIONS:
Procedure: Therapeutic Hypothermia — Participants who are assigned to receive therapeutic hypothermia will be cooled to a target temperature of 33º C plus or minus 1º C (32° to 34º C). This temperature will be maintained for 48 hours (2 days) and then participants will be warmed to a target temperature of 36.75º C plus or minus 0.75º C (36° to 37.5º C). This temperature will be maintained until 120 hours (5 days) after the cardiac arrest.
  Arms: Therapeutic Hypothermia
Procedure: Therapeutic Normothermia — Participants who are assigned to receive therapeutic normothermia will have their temperature maintained at 36.75º C plus or minus 0.75º C (36° to 37.5º C) for 120 hours (5 days) after the cardiac arrest.
  Arms: Therapeutic Normothermia

SUMMARY:
Cardiac arrest is a sudden, unexpected loss of heart function. Therapeutic hypothermia, in which the body's temperature is lowered and maintained several degrees below normal for a period of time, has been used to successfully treat adults who have experienced cardiac arrest. This study will evaluate the efficacy of therapeutic hypothermia at increasing survival rates and reducing the risk of brain injury in infants and children who experience a cardiac arrest while in the hospital.

DETAILED DESCRIPTION:
Cardiac arrest occurs when the heart suddenly stops beating and blood flow to the body is halted. It can occur while people are in the hospital because of a medical condition or while people are out of the hospital as a result of an accident or other cause. Cardiac arrest is a serious event that is associated with high rates of death and long-term disability. When a person experiences cardiac arrest,insufficient amount of blood flow and oxygen can result in brain injury.

Therapeutic hypothermia is a therapy that involves a controlled lowering of the body temperature and then maintenance of this lower temperature for a period of time. Therapeutic hypothermia has been successfully used in adults who experience cardiac arrest to improve survival rates and health outcomes, and it has also been studied in newborn infants who have suffered from perinatal asphyxia. The purpose of this study is to evaluate the efficacy of therapeutic hypothermia at improving survival rates and reducing brain injury in infants and children who experience cardiac arrest while in the hospital.

Study researchers will conduct this study in collaboration with the following two pediatric clinical research networks: the Pediatric Emergency Care Applied Research Network (PECARN), funded by the Emergency Medical Services for Children (EMSC) program, and the National Institute of Child Health and Human Development (NICHD) Collaborative Pediatric Critical Care Research Network (CPCCRN).

The study will enroll infants and children who have suffered a cardiac arrest while in the hospital. Randomization must occur within 6 hours of return of spontaneous circulation. Participants will be randomly assigned to receive either therapeutic hypothermia or therapeutic normothermia. Participants receiving therapeutic hypothermia will have their body temperature reduced to between 32° and 34° Celsius (C) and will remain at this temperature for 2 days. Their body temperature will then be slowly increased to the normal temperature of 36° to 37.5° C, which will be maintained until 5 days after the cardiac arrest. Participants receiving therapeutic normothermia will have their normal temperature maintained between 36° and 37.5° C for 5 days after the cardiac arrest. Special temperature control blankets will be placed to maintain their body temperature in the assigned range. After 5 days, each participant's temperature will be managed by their medical care team.

While participants are in the hospital, they will undergo frequent blood and urine collections, chest x-rays, and temperature measurements; parents of participants will complete questionnaires. When participants are ready to leave the hospital, study researchers will perform a physical and functional assessment. Twenty-eight days after the cardiac arrest, researchers will contact parents of participants to gather information on the participants' health and medical condition. At Months 3 and 12, a child development expert will contact parents to gather medical information. At Month 12, participants will attend a study visit for a neurologic examination and testing with a psychologist trained in rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffered cardiac arrest requiring chest compressions for at least 2 minutes (120 seconds) with ROSC/ROC; AND
* Age greater than 48 hours (with a corrected gestational age of at least 38 weeks) and less than 18 years; AND
* Patient requires continuous mechanical ventilation; AND
* The cardiac arrest was unplanned (i.e., not part of cardiac surgical procedure)

Exclusion Criteria:

* The parent or legal guardian does not speak English or Spanish (the only two languages in which VABS II is standardized)
* Randomization is impossible within six hours of ROSC; OR
* Patient is on extracorporeal membrane oxygenation (ECMO) when arrest occurs; OR
* Continuous infusion of epinephrine or norepinephrine at very high doses (≥2 ug/kg/minute) received immediately prior to randomization; OR Glasgow Coma Scale motor response of five (localizing pain or for infants less than two years, withdraws to touch) or six (obeys commands, or for infants, normal spontaneous movement) prior to randomization; OR
* History of a prior cardiac arrest with chest compressions for at least two minutes during the current hospitalization but outside the 6 hour window for randomization; OR
* Pre-existing terminal illness with life expectancy < 12 months; OR
* Lack of commitment to aggressive intensive care therapies including do not resuscitate orders and other limitations to care; OR
* Cardiac arrest was associated with severe brain, thoracic, or abdominal trauma; OR
* Active and refractory severe bleeding prior to randomization; OR
* Near drowning in ice water with patient core temperature ≤32 °C on presentation; OR
* Patient is pregnant; OR
* Patient participation in a concurrent interventional trial whose protocol, in the judgment of the THAPCA investigators, prevents effective application of one or both THAPCA therapeutic treatment arms, or otherwise significantly interferes with carrying out the THAPCA protocol; OR
* Patient is newborn with acute birth asphyxia; OR

  _ Patient cared for in a neonatal intensive care unit (NICU) after arrest (ie, would not be admitted to PICU); OR
* Patient has sickle cell anemia; OR
* Patient known to have pre-existing cryoglobulinemia; OR
* Central nervous system tumor with ongoing chemotherapy or radiation therapy; OR
* Chronic hypothermia secondary to hypovolemic, pituitary, or related condition for which body temperature is consistently below 37 °C ; OR progressive degenerative encephalopathy; OR
* Any condition in which direct skin surface cooling would be contraindicated, such as large burns, decubitus ulcers, cellulitis, or other conditions with disrupted skin integrity (NOTE: patients with open chest CPR should be included but placement of cooling mattresses will be modified as needed); OR
* Previous enrollment in the THAPCA Trials.

Ages: 48 Hours to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 329 (Actual)
Dates: Start 2009-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Moler, MD, Principal Investigator — University of Michigan; Michael Dean, MD, Principal Investigator — University of Utah
Locations (33):
- United States (25):
  - The Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Loma Linda University Children's Hospital, Loma Linda, California
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - University of California San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Hospital of Atlanta/Emory University, Atlanta, Georgia
  - Riley Children's Hospital, Indianapolis, Indiana
  - Kosair Children's Hospital, Louisville, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Michigan, Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Duke Children's Hospital, Durham, North Carolina
  - Nationwide Children's Hospital in Columbus, Columbus, Ohio
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philidelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - LeBonheur Children's Hospital - University of Tennessee at Memphis, Memphis, Tennessee
  - Children's Medical Center Dallas, Dallas, Texas
  - University of Texas Health Sciences Center of San Antonio, San Antonio, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- The Hospital for Sick Children, Toronto, Ontario, Canada
- United Kingdom (7):
  - Birmingham Children's Hospital, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - University of Hampton, Hampton
  - Alder Hey Children's Hospital, Liverpool
  - Evalina Children's at Guys's and St. Thomas' Hospital, London
  - Great Ormand Street Hospital, London
  - Royal Manchester Children's Hospital, Manchester

REFERENCES:
- [Result] Moler FW, Meert K, Donaldson AE, Nadkarni V, Brilli RJ, Dalton HJ, Clark RS, Shaffner DH, Schleien CL, Statler K, Tieves KS, Hackbarth R, Pretzlaff R, van der Jagt EW, Levy F, Hernan L, Silverstein FS, Dean JM; Pediatric Emergency Care Applied Research Network. In-hospital versus out-of-hospital pediatric cardiac arrest: a multicenter cohort study. Crit Care Med. 2009 Jul;37(7):2259-67. doi: 10.1097/CCM.0b013e3181a00a6a. PMID 19455024
- [Result] Meert KL, Donaldson A, Nadkarni V, Tieves KS, Schleien CL, Brilli RJ, Clark RS, Shaffner DH, Levy F, Statler K, Dalton HJ, van der Jagt EW, Hackbarth R, Pretzlaff R, Hernan L, Dean JM, Moler FW; Pediatric Emergency Care Applied Research Network. Multicenter cohort study of in-hospital pediatric cardiac arrest. Pediatr Crit Care Med. 2009 Sep;10(5):544-53. doi: 10.1097/PCC.0b013e3181a7045c. PMID 19451846
- [Result] Moler FW, Donaldson AE, Meert K, Brilli RJ, Nadkarni V, Shaffner DH, Schleien CL, Clark RS, Dalton HJ, Statler K, Tieves KS, Hackbarth R, Pretzlaff R, van der Jagt EW, Pineda J, Hernan L, Dean JM; Pediatric Emergency Care Applied Research Network. Multicenter cohort study of out-of-hospital pediatric cardiac arrest. Crit Care Med. 2011 Jan;39(1):141-9. doi: 10.1097/CCM.0b013e3181fa3c17. PMID 20935561
- [Result] Moler FW, Silverstein FS, Holubkov R, Slomine BS, Christensen JR, Nadkarni VM, Meert KL, Browning B, Pemberton VL, Page K, Gildea MR, Scholefield BR, Shankaran S, Hutchison JS, Berger JT, Ofori-Amanfo G, Newth CJ, Topjian A, Bennett KS, Koch JD, Pham N, Chanani NK, Pineda JA, Harrison R, Dalton HJ, Alten J, Schleien CL, Goodman DM, Zimmerman JJ, Bhalala US, Schwarz AJ, Porter MB, Shah S, Fink EL, McQuillen P, Wu T, Skellett S, Thomas NJ, Nowak JE, Baines PB, Pappachan J, Mathur M, Lloyd E, van der Jagt EW, Dobyns EL, Meyer MT, Sanders RC Jr, Clark AE, Dean JM; THAPCA Trial Investigators. Therapeutic Hypothermia after In-Hospital Cardiac Arrest in Children. N Engl J Med. 2017 Jan 26;376(4):318-329. doi: 10.1056/NEJMoa1610493. Epub 2017 Jan 24. PMID 28118559
- [Derived] Slomine BS, Silverstein FS, Page K, Holubkov R, Christensen JR, Dean JM, Moler FW; Therapeutic Hypothermia after Pediatric Cardiac Arrest (THAPCA) Trial Investigators. Relationships between three and twelve month outcomes in children enrolled in the therapeutic hypothermia after pediatric cardiac arrest trials. Resuscitation. 2019 Jun;139:329-336. doi: 10.1016/j.resuscitation.2019.03.020. Epub 2019 Mar 26. PMID 30922934
- [Derived] Ichord R, Silverstein FS, Slomine BS, Telford R, Christensen J, Holubkov R, Dean JM, Moler FW; THAPCA Trial Group. Neurologic outcomes in pediatric cardiac arrest survivors enrolled in the THAPCA trials. Neurology. 2018 Jul 10;91(2):e123-e131. doi: 10.1212/WNL.0000000000005773. Epub 2018 Jun 8. PMID 29884735
- [Derived] Slomine BS, Silverstein FS, Christensen JR, Holubkov R, Telford R, Dean JM, Moler FW; Therapeutic Hypothermia after Paediatric Cardiac Arrest (THAPCA) Trial Investigators. Neurobehavioural outcomes in children after In-Hospital cardiac arrest. Resuscitation. 2018 Mar;124:80-89. doi: 10.1016/j.resuscitation.2018.01.002. Epub 2018 Jan 3. PMID 29305927
- [Derived] Holubkov R, Clark AE, Moler FW, Slomine BS, Christensen JR, Silverstein FS, Meert KL, Pollack MM, Dean JM. Efficacy outcome selection in the therapeutic hypothermia after pediatric cardiac arrest trials. Pediatr Crit Care Med. 2015 Jan;16(1):1-10. doi: 10.1097/PCC.0000000000000272. PMID 25268768
- [Derived] Moler FW, Silverstein FS, Meert KL, Clark AE, Holubkov R, Browning B, Slomine BS, Christensen JR, Dean JM. Rationale, timeline, study design, and protocol overview of the therapeutic hypothermia after pediatric cardiac arrest trials. Pediatr Crit Care Med. 2013 Sep;14(7):e304-15. doi: 10.1097/PCC.0b013e31828a863a. PMID 23842585
- [Derived] Pemberton VL, Browning B, Webster A, Dean JM, Moler FW. Therapeutic hypothermia after pediatric cardiac arrest trials: the vanguard phase experience and implications for other trials. Pediatr Crit Care Med. 2013 Jan;14(1):19-26. doi: 10.1097/PCC.0b013e31825b860b. PMID 23295834
- See also: IH THAPCA Abstract — https://www.ncbi.nlm.nih.gov/pubmed/28118559

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Therapeutic Hypothermia | Therapeutic Normothermia
Started | 166 (Among the 166 Started, 161 received Therapeutic Hypothermia and 5 received no treatment.) | 163 (Among the 163 Started, 160 received Therapeutic Normothermia and 3 received no treatment.)
Completed | 166 (1-year vital status available for all 166 Started patients.) | 161 (Of 161 with 1-year vital status, 158 had received Therapeutic Normothermia, 3 received no treatment.)
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Therapeutic Hypothermia | Therapeutic Normothermia | Total
Number analyzed (Participants) | 166 | 163 | 329
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 1.4 [0.3 to 5.7] | 0.6 [0.2 to 6.3] | 1.0 [0.2 to 5.8]
Age, Customized [Count of Participants; unit: Participants]
  Age Category: < 2 yr | 97 | 104 | 201
  Age Category: 2 - <12 yr | 48 | 35 | 83
  Age Category: 12 - 17 yr | 21 | 24 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 64 | 133
  Male | 97 | 99 | 196

OUTCOME MEASURES:

1. Primary Outcome: Survival With Good Neurobehavioral Outcome
Description: Survival at one-year anniversary of cardiac arrest, with a standardized VABS-II score of 70 or greater per evaluation performed at any time from 30 days prior to until 183 days after the one-year anniversary of cardiac arrest. Higher values of VABS-II represent a better outcome.
Time Frame: Survival was assessed at one-year anniversary of cardiac arrest; among survivors at this one-year anniversary, the VABS-II valid assessment window ranged from 30 days prior to until 183 days after the one-year anniversary date.
Population: Subjects with baseline VABS-II >= 70, OR unavailable baseline VABS-II but Pediatric Overall Performance Category (POPC) score and Pediatric Cerebral Overall Performance Category (PCPC) both reflecting none or mild disability (1 or 2), are eligible for the primary analysis. Population is analysis-eligible patients with available primary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Hypothermia | Therapeutic Normothermia
Number analyzed (Participants) | 133 | 124
Participants
  Alive with VABS-II >=70 at 1 year | 48 | 48
  Died or Alive with VABS-II <70 at 1 year | 85 | 76
Statistical Analysis 1: Comparison: Therapeutic Hypothermia vs Therapeutic Normothermia; Test type: Superiority; p = 0.63, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test was used adjusting for age category at time of randomization (<2 years, 2 to <12 years, or >=12 years); Risk Difference (RD) = -2.6, 95% CI 2-sided [-14.5 to 9.2]

2. Secondary Outcome: Survival
Description: Survival at one year after cardiac arrest
Time Frame: Measured at one-year anniversary of cardiac arrest.
Population: All randomized patients with available vital status (alive or deceased) at one year after cardiac arrest.
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Hypothermia | Therapeutic Normothermia
Number analyzed (Participants) | 166 | 161
Participants
  Alive at 1 year | 81 | 74
  Died at 1 year | 85 | 87
Statistical Analysis 1: Comparison: Therapeutic Hypothermia vs Therapeutic Normothermia; Test type: Superiority; p = 0.56, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 2.8, 95% CI 2-sided [-8.0 to 13.7]

3. Secondary Outcome: Change in Neurobehavioral Function From Pre-cardiac Arrest to 12 Months Post-cardiac Arrest
Description: Change in VABS-II score from baseline to one year, with death at 1 year treated as worst possible outcome, and lowest possible VABS-II score at one year (regardless of baseline VABS-II score) treated as the second worst possible outcome. Since higher levels of VABS-II represent a better outcome, a larger decline (large negative magnitude of change) in VABS-II score from baseline to one year represents a worse outcome.
Time Frame: as for outcome 1
Population: All randomized subjects with available data for this outcome (this implies a child must be either dead at 1 year, have the lowest possible value for the VABS-II score at 1 year, or if neither of these two criteria applies, must have both baseline VABS-II and 1-year VABS-II scores available to allow calculation of change in VABS-II score)
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Hypothermia | Therapeutic Normothermia
Number analyzed (Participants) | 164 | 153
Participants
  Dead at 1 year | 85 | 87
  Lowest possible VABS-II at 1 year | 1 | 0
  1-year decrease in VABS-II >30 points | 12 | 8
  1-year decrease in VABS-II 16-30 points | 17 | 14
  1-year decrease in VABS-II <=15 points or improved | 49 | 44
Statistical Analysis 1: Comparison: Therapeutic Hypothermia vs Therapeutic Normothermia; Test type: Superiority; p = 0.70, Stratified Mann-Whitney Test; Test stratified by age category (<2 years, 2 to <12 years, or >=12 years), for continuous (NOT categorized as reported above) 1-year change in VABS-II; As the (nonparametric) comparison treated 1-year deaths as worst possible outcomes and worst possible 1-year VABS-II as next worst possible outcomes, using change in VABS-II for other participants alive at 1 year, no relevant estimation of effect size is possible for this secondary outcome

4. Secondary Outcome: Neuropsychological Scores (for Participants Who Survive)
Description: Functioning, as assessed by the Mullen Early Learning Composite (for children age < 5 years 9 months) or by the 2-subset version of the Wechsler Abbreviated Scale of Intelligence (WASI). As these two function measures are scaled in the same fashion, the two age groups are combined.
Time Frame: Measured at Month 12
Population: Randomized children alive at one year with neuropsychological score available.
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Hypothermia | Therapeutic Normothermia
Number analyzed (Participants) | 68 | 48
Participants
  Lowest possible score | 18 | 8
  <70 (well below average) | 18 | 11
  70 - 84 (below average) | 9 | 14
  85-115 (average) | 21 | 13
  >115 (above average) | 2 | 2
Statistical Analysis 1: Comparison: Therapeutic Hypothermia vs Therapeutic Normothermia; Test type: Superiority; p = 0.46, Wilcoxon (Mann-Whitney); Test used the continuous (NOT categorized as reported above) neuropsychological scores, with "Lowest Possible Score" treated as lowest possible value

5. Other Pre Specified Outcome: Neurological Abnormality Scores (for Participants Who Survive)
Time Frame: Measured at Month 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: For all-cause mortality, results reflect vital status at 12 months. Serious adverse events and other (not serious) adverse events were collected for 14 days after treatment was initiated.
Description: For adverse events, denominators reflect Safety Population of patients receiving each treatment: 161 patients receiving Therapeutic Hypothermia and 160 patients receiving Therapeutic Normothermia. However, for all-cause mortality at 12 months, denominators can only include those with known 12-month vital status. Since 2 participants who received Therapeutic Normothermia were lost to follow-up at 1 year, the Therapeutic Normothermia denominator for all-cause mortality is 158 rather than 160.
Arm/Group | Therapeutic Hypothermia | Therapeutic Normothermia
All-Cause Mortality (participants affected / at risk) | 82/161 | 84/158
Serious Adverse Events (participants affected / at risk) | 85/161 | 91/160
Other Adverse Events (participants affected / at risk) | 151/161 | 146/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapeutic Hypothermia (N=161) | Therapeutic Normothermia (N=160)
Coagulopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
DIC (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypercoagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arrest cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial perforation (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (3) | 4 (4)
Cardiac arrest (Cardiac disorders) | 18 (20) | 16 (17)
Cardiac failure (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac insufficiency (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac ischemia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 1 (1)
Cardiopulmonary arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 2 (2)
Dysrhythmias (Cardiac disorders) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Recurrent ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Bowel perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hemorrhage intraabdominal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ischemia bowel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Necrotizing enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Brain death (General disorders) | 1 (1) | 0 (0)
Catheter site bleeding (General disorders) | 2 (2) | 0 (0)
Clotting of extracorporeal circuit (General disorders) | 0 (0) | 1 (1)
Extracorporeal membrane oxygenation complication (General disorders) | 1 (1) | 1 (1)
Multi organ failure (General disorders) | 1 (1) | 1 (1)
Multi-organ failure (General disorders) | 2 (2) | 1 (1)
Multiple organ failure (General disorders) | 2 (2) | 3 (3)
Bacterial tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella pneumoniae infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Respiratory infection (Infections and infestations) | 2 (2) | 2 (3)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 2 (2)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 2 (2)
Acute subdural hematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Brain herniation (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Epidural hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration of lung with open wound into thorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Atrial pressure increased (Investigations) | 1 (1) | 0 (0)
Blood culture positive (Investigations) | 0 (0) | 2 (2)
Cardiac output decreased (Investigations) | 1 (1) | 1 (1)
HIE (Investigations) | 0 (0) | 1 (1)
Sputum culture positive (Investigations) | 1 (1) | 0 (0)
Acidosis aggravated (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Anoxic brain damage (Nervous system disorders) | 5 (5) | 8 (8)
Anoxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral edema (Nervous system disorders) | 2 (2) | 3 (3)
Cerebral infarct (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischemia (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Hemorrhagic transformation stroke (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxic brain damage (Nervous system disorders) | 3 (3) | 2 (2)
Hypoxic encephalopathy (Nervous system disorders) | 6 (6) | 6 (6)
Intracerebral hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 2 (2) | 1 (1)
Intraventricular hemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Ischemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Middle cerebral artery infarct (Nervous system disorders) | 1 (1) | 0 (0)
Middle cerebral artery stroke (Nervous system disorders) | 0 (0) | 1 (1)
Neurological status deterioration (Nervous system disorders) | 1 (1) | 0 (0)
Reflexes absent (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 3 (3) | 0 (0)
Subarachnoid hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1) | 4 (4)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Embolism pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary hypertension aggravated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thoracic hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Aortic rupture (Vascular disorders) | 0 (0) | 1 (1)
Critical limb ischemia (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 4 (4) | 2 (2)
Hypotension aggravated (Vascular disorders) | 3 (3) | 0 (0)
Ischemia (Vascular disorders) | 2 (2) | 1 (1)
Ischemia peripheral (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapeutic Hypothermia (N=161) | Therapeutic Normothermia (N=160)
Anemia (Blood and lymphatic system disorders) | 10 (10) | 9 (9)
Coagulopathy (Blood and lymphatic system disorders) | 10 (10) | 13 (13)
DIC (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Hemolysis (Blood and lymphatic system disorders) | 4 (4) | 3 (3)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypercoagulation (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 5 (5) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Methemoglobinemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Monocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (12) | 10 (10)
Thrombocytopenia aggravated (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
AV nodal tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Accelerated idioventricular rhythm (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 2 (2)
Atrial bigeminy (Cardiac disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 2 (2) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Bradycardia (Cardiac disorders) | 15 (16) | 5 (5)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Congestive cardiac failure aggravated (Cardiac disorders) | 1 (1) | 0 (0)
Cyanosis (Cardiac disorders) | 1 (1) | 0 (0)
Cyanosis peripheral (Cardiac disorders) | 0 (0) | 1 (1)
Ectopic atrial beats (Cardiac disorders) | 1 (1) | 0 (0)
Effusion pericardial (Cardiac disorders) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Heart block (Cardiac disorders) | 1 (1) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Junctional rhythm (Cardiac disorders) | 3 (3) | 1 (1)
Junctional tachycardia (Cardiac disorders) | 3 (3) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular hypokinesia (Cardiac disorders) | 1 (1) | 0 (0)
Monomorphic ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial depression (Cardiac disorders) | 0 (0) | 1 (1)
PVC's (Cardiac disorders) | 3 (4) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2) | 2 (2)
Premature atrial contraction (Cardiac disorders) | 0 (0) | 1 (1)
Premature ventricular contractions (Cardiac disorders) | 0 (0) | 1 (1)
Right bundle branch block (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
SVT (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Tachycardia (Cardiac disorders) | 3 (3) | 6 (7)
Trigeminy (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular ectopics (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 7 (9)
Antithrombin III deficiency (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Methylenetetrahydrofolate reductase deficiency (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Thyroglossal duct cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 3 (3) | 4 (4)
Adrenal mass (Endocrine disorders) | 1 (1) | 0 (0)
Diabetes insipidus (Endocrine disorders) | 3 (3) | 5 (5)
Eye movement disorder (Eye disorders) | 0 (0) | 2 (2)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1)
Fixed dilated pupils (Eye disorders) | 0 (0) | 1 (1)
Fixed pupils (Eye disorders) | 1 (1) | 1 (1)
Scleral edema (Eye disorders) | 1 (1) | 0 (0)
Abdominal compartment syndrome (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Absent bowel sounds (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 9 (9) | 9 (9)
Bleeding esophageal varices (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blood stool (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bloody diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bloody stool (Gastrointestinal disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Distended abdomen (Gastrointestinal disorders) | 1 (1) | 1 (1)
Distended bowel (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Emesis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 2 (2)
Ileus of bowel (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Loose stools (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric edema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Necrotizing enterocolitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral lesion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic insufficiency (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 4 (4)
Perihepatic fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Swelling of tongue (Gastrointestinal disorders) | 0 (0) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
UGI bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ulcer lip (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anasarca (General disorders) | 5 (5) | 8 (8)
Catheter site bleeding (General disorders) | 11 (12) | 9 (9)
Catheter site hemorrhage (General disorders) | 0 (0) | 1 (1)
Clotting of extracorporeal circuit (General disorders) | 3 (3) | 3 (3)
Dependent edema (General disorders) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 1 (1) | 1 (1)
Edema (General disorders) | 4 (4) | 2 (2)
Edema aggravated (General disorders) | 1 (1) | 1 (1)
Edema generalized (General disorders) | 0 (0) | 1 (1)
Edema trunk (General disorders) | 1 (1) | 1 (1)
Edematous weight gain (General disorders) | 0 (0) | 1 (1)
Extracorporeal membrane oxygenation complication (General disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 10 (13) | 11 (11)
Generalized edema (General disorders) | 0 (0) | 2 (2)
Hyperthermia (General disorders) | 3 (4) | 3 (3)
Hypothermia (General disorders) | 2 (2) | 2 (2)
Infusion site infiltration (General disorders) | 0 (0) | 1 (2)
Intermittent fever (General disorders) | 1 (1) | 0 (0)
Multiple organ failure (General disorders) | 1 (1) | 0 (0)
Necrosis (General disorders) | 0 (0) | 1 (1)
Needle stick/puncture (General disorders) | 1 (1) | 0 (0)
Opiate withdrawal symptoms (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1)
Peripheral edema (General disorders) | 0 (0) | 1 (1)
Pitting edema (General disorders) | 0 (0) | 1 (1)
Pyrexial (General disorders) | 0 (0) | 1 (1)
Shivering (General disorders) | 5 (5) | 1 (1)
Swelling (General disorders) | 1 (1) | 0 (0)
Swelling arm (General disorders) | 0 (0) | 1 (1)
Swelling of legs (General disorders) | 1 (1) | 1 (1)
Swelling of limb (General disorders) | 1 (1) | 1 (1)
Weakness generalized (General disorders) | 0 (0) | 1 (1)
Acute liver failure (Hepatobiliary disorders) | 2 (2) | 0 (0)
Function liver abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Function liver decreased (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic insufficiency (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic ischemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic shock (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 2 (2) | 2 (2)
Hepatopathy (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatosplenomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 3 (3) | 6 (6)
Ischemic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hypogammaglobulinemia (Immune system disorders) | 0 (0) | 2 (2)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Abscess hand (Infections and infestations) | 1 (1) | 0 (0)
Bacterial eye infection (Infections and infestations) | 1 (1) | 0 (0)
Bacterial infection due to staphylococcus aureus (Infections and infestations) | 1 (1) | 1 (1)
Bacterial tracheitis (Infections and infestations) | 2 (2) | 1 (1)
Candida albicans infection (Infections and infestations) | 1 (1) | 0 (0)
Cardiac valve vegetation (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Escherichia coli infection (Infections and infestations) | 0 (0) | 2 (2)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Eye infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Eye infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Fungal rash (Infections and infestations) | 2 (2) | 0 (0)
Fungemia (Infections and infestations) | 1 (1) | 0 (0)
Gram-positive bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Herpetic stomatitis (Infections and infestations) | 0 (0) | 1 (1)
Infection MRSA (Infections and infestations) | 0 (0) | 1 (1)
Infection pseudomonas aeruginosa (Infections and infestations) | 1 (1) | 0 (0)
Infection respiratory (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
MRSA wound infection (Infections and infestations) | 0 (0) | 1 (1)
Parvovirus B19 infection (Infections and infestations) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pleural infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 1 (1)
Pneumonia due to Escherichia coli (E. Coli) (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory infection (Infections and infestations) | 3 (4) | 10 (10)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 4 (4) | 3 (3)
Sepsis (Infections and infestations) | 4 (4) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Sinus infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Streptococcus pneumoniae pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Thrush (Infections and infestations) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1) | 1 (1)
UTI (Infections and infestations) | 1 (1) | 1 (1)
Urinary infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (5) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection fungal (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Ventilator associated pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Abrasions (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Bloody airway discharge (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Bronchial injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bruise (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Collapse of lung (Injury, poisoning and procedural complications) | 7 (7) | 1 (1)
Ear injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Endotracheal reintubation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Foot injury (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Injury to kidney (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Knee injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laryngeal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nerve damage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Operation site bleed (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative bleeding (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radial artery injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Shunt thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Unintended endotracheal extubation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound oozing (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ALT increased (Investigations) | 7 (7) | 3 (3)
APTT increased (Investigations) | 1 (1) | 1 (1)
APTT prolonged (Investigations) | 3 (3) | 0 (0)
AST increased (Investigations) | 5 (5) | 5 (5)
Abnormal EEG (Investigations) | 3 (3) | 1 (1)
Adenovirus test positive (Investigations) | 1 (1) | 0 (0)
Albumin decreased (Investigations) | 1 (1) | 0 (0)
Albumin low (Investigations) | 1 (1) | 1 (1)
Ammonia increased (Investigations) | 0 (0) | 1 (1)
Amylase high (Investigations) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 5 (5) | 4 (4)
Antithrombin III decreased (Investigations) | 2 (2) | 4 (4)
Antithrombin III increased (Investigations) | 0 (0) | 1 (1)
Arterial blood pH decreased (Investigations) | 0 (0) | 1 (1)
Arterial catheterisation abnormal (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Atrial pressure increased (Investigations) | 1 (1) | 0 (0)
B-type natriuretic peptide (Investigations) | 0 (0) | 1 (1)
BNP increased (Investigations) | 1 (1) | 2 (2)
BUN increased (Investigations) | 2 (2) | 6 (6)
Bacteria sputum identified (Investigations) | 1 (2) | 0 (0)
Bacteria stool identified (Investigations) | 0 (0) | 1 (1)
Bacteria urine identified (Investigations) | 1 (1) | 0 (0)
Band neutrophil count increased (Investigations) | 1 (1) | 3 (3)
Base excess abnormal (Investigations) | 0 (0) | 1 (1)
Base excess decreased (Investigations) | 1 (1) | 0 (0)
Base excess increased (Investigations) | 0 (0) | 2 (2)
Bilirubin elevated (Investigations) | 1 (1) | 0 (0)
Bilirubin increased (Investigations) | 6 (6) | 3 (3)
Blood LDH abnormal (Investigations) | 0 (0) | 1 (1)
Blood amylase increased (Investigations) | 0 (0) | 1 (1)
Blood bicarbonate decreased (Investigations) | 3 (3) | 0 (0)
Blood bicarbonate increased (Investigations) | 1 (1) | 1 (1)
Blood bicarbonate low (Investigations) | 0 (0) | 1 (1)
Blood bilirubin decreased (Investigations) | 0 (0) | 1 (1)
Blood culture positive (Investigations) | 5 (6) | 6 (7)
Blood lactic acid increased (Investigations) | 1 (1) | 0 (0)
Blood phosphorus increased (Investigations) | 3 (3) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Blood pressure diastolic low (Investigations) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1)
Blood urea nitrogen increased (Investigations) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 1 (1)
Brain natriuretic peptide abnormal (Investigations) | 0 (0) | 1 (1)
Brain natriuretic peptide increased (Investigations) | 1 (1) | 3 (3)
C-reactive protein abnormal (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 3 (3) | 1 (1)
CK increased (Investigations) | 2 (2) | 0 (0)
CPK increased (Investigations) | 1 (1) | 1 (2)
CRP increased (Investigations) | 3 (3) | 1 (1)
Calcium ionized increased (Investigations) | 1 (1) | 0 (0)
Calcium low (Investigations) | 1 (1) | 3 (3)
Capillary nail refill test abnormal (Investigations) | 1 (1) | 0 (0)
Carbon dioxide decreased (Investigations) | 0 (0) | 1 (1)
Carbon dioxide increased (Investigations) | 0 (0) | 1 (1)
Carbon dioxide total decreased (Investigations) | 1 (1) | 0 (0)
Carbon dioxide total increased (Investigations) | 0 (0) | 1 (1)
Cardiac enzymes increased (Investigations) | 2 (2) | 0 (0)
Cardiac output decreased (Investigations) | 2 (2) | 3 (3)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1)
Casts urinary granular (Investigations) | 2 (2) | 0 (0)
Central venous pressure decreased (Investigations) | 0 (0) | 1 (1)
Central venous pressure increased (Investigations) | 0 (0) | 1 (1)
Chloride decreased (Investigations) | 1 (1) | 0 (0)
Chloride low (Investigations) | 1 (1) | 1 (1)
Clotting time increased (Investigations) | 1 (1) | 0 (0)
Coagulation factor II level decreased (Investigations) | 1 (1) | 0 (0)
Coronavirus test positive (Investigations) | 1 (1) | 0 (0)
Creatine kinase increased (Investigations) | 0 (0) | 1 (1)
Creatinine high (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 2 (2) | 6 (6)
Culture throat positive (Investigations) | 1 (1) | 0 (0)
Culture wound positive (Investigations) | 1 (1) | 0 (0)
Decreased hemoglobin (Investigations) | 0 (0) | 4 (4)
Drug level in blood increased (Investigations) | 1 (1) | 0 (0)
EEG abnormal (Investigations) | 3 (3) | 0 (0)
Elevated liver enzymes (Investigations) | 3 (3) | 0 (0)
Fecal occult blood positive (Investigations) | 0 (0) | 1 (1)
Fibrin D dimer increased (Investigations) | 4 (4) | 0 (0)
Fibrinogen decreased (Investigations) | 7 (7) | 2 (2)
Fibrinogen increased (Investigations) | 3 (3) | 0 (0)
Free hemoglobin present (Investigations) | 0 (0) | 1 (1)
Free plasma hemoglobin (Investigations) | 1 (1) | 0 (0)
Glucose decreased (Investigations) | 0 (0) | 2 (2)
Glucose high (Investigations) | 1 (1) | 1 (1)
Glucose increased (Investigations) | 2 (2) | 4 (4)
HIV positive (Investigations) | 1 (1) | 0 (0)
Haemoglobin abnormal (Investigations) | 0 (0) | 1 (1)
Haemoglobin low (Investigations) | 4 (4) | 1 (1)
Heart rate low (Investigations) | 0 (0) | 1 (1)
Hematocrit decreased (Investigations) | 0 (0) | 1 (1)
Hematocrit low (Investigations) | 2 (2) | 1 (1)
Hemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Hemoglobin increased (Investigations) | 1 (1) | 2 (2)
INR decreased (Investigations) | 0 (0) | 1 (2)
INR increased (Investigations) | 1 (1) | 2 (2)
Increased platelets (Investigations) | 2 (2) | 0 (0)
Increased serum creatinine (Investigations) | 0 (0) | 1 (1)
Ionized calcium decreased (Investigations) | 2 (2) | 7 (7)
Ionized calcium increased (Investigations) | 2 (2) | 0 (0)
LDH decreased (Investigations) | 0 (0) | 2 (2)
LDH increased (Investigations) | 3 (3) | 3 (3)
LFTs raised (Investigations) | 0 (0) | 1 (1)
Lactate blood increased (Investigations) | 0 (0) | 1 (1)
Lactate dehydrogenase (Investigations) | 0 (0) | 1 (1)
Lactate dehydrogenase increased (Investigations) | 13 (13) | 5 (5)
Lactate increased (Investigations) | 3 (3) | 1 (1)
Lipase increased (Investigations) | 9 (9) | 5 (5)
Liver enzyme abnormal (Investigations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1)
Liver function tests raised (Investigations) | 1 (1) | 3 (3)
Long QT (Investigations) | 1 (1) | 0 (0)
Low pH (Investigations) | 3 (3) | 1 (1)
Low platelets (Investigations) | 6 (7) | 3 (3)
Lung function abnormal (Investigations) | 0 (0) | 1 (1)
Magnesium decreased (Investigations) | 5 (5) | 5 (5)
Magnesium increased (Investigations) | 1 (1) | 0 (0)
Magnesium low (Investigations) | 2 (2) | 1 (1)
Mean arterial pressure increased (Investigations) | 1 (2) | 1 (1)
Methicillin-resistant Staphylococcus aureus test positive (Investigations) | 0 (0) | 2 (2)
Mycoplasma antibody positive (Investigations) | 0 (0) | 1 (1)
Neutrophil count low (Investigations) | 1 (1) | 0 (0)
Nonspecific ST segment change (Investigations) | 2 (2) | 0 (0)
Occult blood positive (Investigations) | 1 (1) | 1 (1)
Osmolality increased (Investigations) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 4 (5) | 12 (12)
PCO2 abnormal (Investigations) | 0 (0) | 1 (1)
PCO2 decreased (Investigations) | 1 (1) | 1 (1)
PCO2 elevated (Investigations) | 2 (2) | 3 (4)
PO2 decreased (Investigations) | 0 (0) | 2 (6)
PT increased (Investigations) | 0 (0) | 1 (1)
PT prolonged (Investigations) | 0 (0) | 1 (1)
PTT prolonged (Investigations) | 0 (0) | 1 (1)
Pancreatic enzymes increased (Investigations) | 1 (1) | 3 (3)
Peripheral pulse decreased (Investigations) | 1 (1) | 0 (0)
Phosphate high (Investigations) | 2 (2) | 0 (0)
Phosphate increased (Investigations) | 2 (2) | 1 (1)
Phosphate low (Investigations) | 2 (3) | 0 (0)
Phosphorus low (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Platelets decreased (Investigations) | 1 (1) | 2 (2)
Potassium decreased (Investigations) | 4 (5) | 2 (2)
Potassium high (Investigations) | 1 (1) | 0 (0)
Potassium increased (Investigations) | 1 (1) | 1 (1)
Potassium low (Investigations) | 0 (0) | 1 (1)
Prealbumin decreased (Investigations) | 0 (0) | 1 (1)
Procalcitonin increased (Investigations) | 0 (0) | 1 (1)
Protein total decreased (Investigations) | 0 (0) | 1 (1)
Prothrombin time increased (Investigations) | 1 (1) | 1 (1)
Pulse absent (Investigations) | 1 (1) | 0 (0)
Pulse pressure abnormal (Investigations) | 0 (0) | 1 (1)
QRS widened (Investigations) | 1 (1) | 0 (0)
QT interval prolonged (Investigations) | 1 (1) | 0 (0)
RBC decreased (Investigations) | 0 (0) | 1 (1)
RDW increased (Investigations) | 0 (0) | 1 (1)
Raised LFTs (Investigations) | 0 (0) | 2 (2)
Right atrial pressure increased (Investigations) | 0 (0) | 1 (1)
SGOT increased (Investigations) | 1 (1) | 0 (0)
ST segment elevation (Investigations) | 1 (1) | 0 (0)
Serum serotonin decreased (Investigations) | 1 (1) | 0 (0)
Serum sodium decreased (Investigations) | 0 (0) | 1 (1)
Sodium increased (Investigations) | 4 (4) | 1 (1)
Sputum culture positive (Investigations) | 15 (16) | 11 (12)
Stool Guaiac test positive (Investigations) | 0 (0) | 1 (1)
Thyroid stimulating hormone decreased (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 2 (2) | 0 (0)
Transaminitis (Investigations) | 4 (4) | 3 (3)
Tri-iodothyronine low (Investigations) | 1 (1) | 0 (0)
Triglyceride increased (Investigations) | 1 (1) | 2 (2)
Triglycerides high (Investigations) | 0 (0) | 1 (1)
Troponin I increased (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 7 (7) | 2 (2)
Urea increased (Investigations) | 1 (2) | 1 (1)
Urea nitrogen increased (Investigations) | 1 (1) | 0 (0)
Urine culture positive (Investigations) | 8 (8) | 6 (7)
Urine output decreased (Investigations) | 7 (7) | 5 (5)
Urine output increased (Investigations) | 3 (3) | 1 (1)
VEP's abnormal (Investigations) | 0 (0) | 1 (1)
Vascular resistance pulmonary increased (Investigations) | 1 (1) | 0 (0)
Venous blood pH decreased (Investigations) | 0 (0) | 1 (1)
Venous oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
Viral test positive (Investigations) | 0 (0) | 1 (1)
Viral titer increased (Investigations) | 1 (1) | 0 (0)
WBC decreased (Investigations) | 2 (2) | 4 (4)
WBC increased (Investigations) | 3 (3) | 2 (2)
White blood cell agglutination present (Investigations) | 2 (2) | 0 (0)
White blood cell count high (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 2 (2) | 5 (5)
White blood cell increased (Investigations) | 0 (0) | 1 (1)
pH increased (Investigations) | 2 (4) | 3 (3)
Acidemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Acidosis aggravated (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acidosis metabolic (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Cerebral salt-wasting syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Fluid imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperammonemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperamylasemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperchloremia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 21 (21) | 20 (20)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3) | 6 (6)
Hyperlactatemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 8 (8) | 7 (7)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 17 (17) | 11 (11)
Hypochloremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 8 (8) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 44 (52) | 31 (33)
Hypomagnesemia (Metabolism and nutrition disorders) | 10 (10) | 10 (10)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 6 (6) | 4 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 10 (10) | 7 (7)
Hypoproteinemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypovolemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Lactic acidosis (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 5 (6) | 4 (4)
Metabolic alkalosis (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Volume overload (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Weakness in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Anoxic brain damage (Nervous system disorders) | 3 (3) | 1 (1)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral dysfunction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral edema (Nervous system disorders) | 1 (1) | 3 (3)
Cerebral hemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral infarct (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral ischemia (Nervous system disorders) | 1 (1) | 0 (0)
Choreiform (Nervous system disorders) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Convulsive movements (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 3 (3) | 1 (1)
Encephalopathy acute (Nervous system disorders) | 1 (1) | 0 (0)
Focal seizures (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Hemorrhage cerebral (Nervous system disorders) | 1 (1) | 0 (0)
Hypertonia (Nervous system disorders) | 0 (0) | 1 (1)
Hypertonicity (Nervous system disorders) | 0 (0) | 1 (1)
Hypotonia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxic brain damage (Nervous system disorders) | 2 (2) | 0 (0)
Hypoxic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Increased intracranial pressure (Nervous system disorders) | 1 (1) | 0 (0)
Infarct cerebral (Nervous system disorders) | 0 (0) | 1 (1)
Intracerebral bleed (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 4 (4)
Intraventricular hemorrhage (Nervous system disorders) | 0 (0) | 2 (2)
Ischemia cerebral (Nervous system disorders) | 1 (1) | 0 (0)
Middle cerebral artery infarct (Nervous system disorders) | 1 (1) | 0 (0)
Movements involuntary of limbs (Nervous system disorders) | 1 (1) | 0 (0)
Movements reduced (Nervous system disorders) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1)
Neurological status deterioration (Nervous system disorders) | 0 (0) | 1 (1)
Paresis (Nervous system disorders) | 0 (0) | 1 (1)
Periventricular leukomalacia (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 16 (17) | 10 (10)
Seizures (Nervous system disorders) | 12 (13) | 16 (17)
Stroke (Nervous system disorders) | 2 (2) | 1 (1)
Subarachnoid hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Subependymal hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Thalamic syndrome (Nervous system disorders) | 3 (3) | 1 (1)
Tonic clonic movements (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Unresponsive (Nervous system disorders) | 1 (1) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 2 (2) | 0 (0)
Weakness left or right side (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 4 (4) | 6 (6)
Agitation aggravated (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety aggravated (Psychiatric disorders) | 0 (0) | 1 (1)
Disorientated (Psychiatric disorders) | 0 (0) | 1 (1)
Drug dependence (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 1 (1)
Increased agitation (Psychiatric disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 4 (4)
Acute renal failure (Renal and urinary disorders) | 4 (4) | 1 (1)
Acute renal insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0)
Anuria (Renal and urinary disorders) | 3 (3) | 1 (1)
Azotemia (Renal and urinary disorders) | 1 (1) | 1 (1)
Bladder distension (Renal and urinary disorders) | 1 (1) | 0 (0)
Bleeding urogenital (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2) | 3 (3)
Hematuria aggravated (Renal and urinary disorders) | 0 (0) | 1 (1)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Oliguria (Renal and urinary disorders) | 2 (2) | 2 (2)
Renal disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 5 (5) | 2 (2)
Renal failure aggravated (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal function abnormal (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal function disorder (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal insufficiency (Renal and urinary disorders) | 2 (2) | 3 (3)
Uremia (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Genital rash (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Paraphimosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic fluid collection (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Priapism (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Scrotal edema (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute on chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 17 (20)
Bronchial hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypercarbia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hyperoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Increased work of breathing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Labored breathing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Lobar collapse (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Lung hyperinflation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Mediastinal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Necrosis of bronchioli (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nose bleed (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 18 (21) | 17 (21)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 11 (13)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (8)
Pulmonary edema aggravated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 5 (5)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary pneumatocele (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary vascular disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary venous congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Respiratory failure aggravated (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sputum bloody (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Tension pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Bed sore (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (3) | 3 (3)
Blistering (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Blisters (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Blood blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bullae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bullous lesions (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Contact dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hives (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Mottled skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pressure sore (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (3)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash over arms (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash trunk (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Redness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin breakdown (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Extracorporeal membrane oxygenation (Surgical and medical procedures) | 1 (1) | 0 (0)
Extubation (Surgical and medical procedures) | 0 (0) | 1 (2)
Pulmonary artery banding (Surgical and medical procedures) | 0 (0) | 1 (1)
Thoracic cavity drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Acute hypotension (Vascular disorders) | 1 (1) | 0 (0)
Aortic thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Arterial thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Axillary vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Bleeding (Vascular disorders) | 6 (6) | 12 (14)
Blood pressure high (Vascular disorders) | 0 (0) | 1 (2)
Blood pressure labile (Vascular disorders) | 0 (0) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 1 (1) | 3 (3)
Clot blood (Vascular disorders) | 0 (0) | 1 (1)
Cold extremities (Vascular disorders) | 0 (0) | 1 (1)
DVT of legs (Vascular disorders) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Deep vein thrombosis leg (Vascular disorders) | 0 (0) | 1 (1)
Deep venous thrombosis femoral (Vascular disorders) | 1 (1) | 1 (1)
Digital necrosis (Vascular disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 1 (1)
Embolus upper extremity (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Femoral artery thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hemodynamic instability (Vascular disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 18 (19) | 14 (14)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypoperfusion (Vascular disorders) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 26 (32) | 24 (26)
Hypotension aggravated (Vascular disorders) | 4 (4) | 4 (4)
Hypotensive episode (Vascular disorders) | 1 (1) | 0 (0)
Inferior venacaval thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Ischemia (Vascular disorders) | 0 (0) | 1 (1)
Ischemia peripheral (Vascular disorders) | 4 (4) | 1 (1)
Jugular vein distension (Vascular disorders) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Leg ischemia (Vascular disorders) | 1 (1) | 0 (0)
Low BP (Vascular disorders) | 0 (0) | 2 (2)
Low blood pressure (Vascular disorders) | 1 (1) | 1 (1)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Poor peripheral perfusion (Vascular disorders) | 2 (2) | 7 (7)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)
Superior venacaval thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis vena cava inferior (Vascular disorders) | 1 (1) | 0 (0)
Venous insufficiency (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No